CLINICAL TRIAL: NCT01029977
Title: Imaging Modality Effects on the Multi-dimensional InfraRed Analysis (MIRA) Technology
Status: Withdrawn | Type: Observational
Why Stopped: Re-definition of MIRA technology goals.
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 960-PRL-002
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2015-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effect of everyday practice modalities (mammography, US) on the MIRA technology.

DETAILED DESCRIPTION:
The objective of the current clinical study is to collect sufficient MIRA imaging data of subjects arriving for a routine screening mammography, before and after they undergo the mammography. This is in order to reach a conclusion whether the the firm breast compression involved in the mammography procedure affects the performance of the MIRA technology. At the current stage of the development of the device, the goal of this clinical trial is in no way to arrive at a statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Gender: female
* Age: 50 years and older
* Subjects summoned for a routine screening mammography, ultrasound, diagnostic mammography or breast biopsy.
* Subject who have signed an informed consent form.

Exclusion Criteria:

* Subjects who have had a mammography, ultrasound, and/or MRI examination performed on the day of the study, PRIOR to their FIRST imaging session with the RealImager.
* Subjects who have undergone any type of breast surgery throughout the 6 weeks preceding the study.
* Subjects who have had a breast biopsy performed throughout the 6 weeks preceding the study.
* Subjects who have undergone a mastectomy.
* Subjects who have undergone a lumpectomy.
* Subjects who have a large scar (causing breast deformation).
* Subjects who have previously undergone or are currently undergoing breast radiation therapy.
* Subjects who have previously undergone or are currently undergoing chemotherapy.
* Subjects with prior breast reduction surgery or breast augmentation surgery.
* Subjects who are pregnant.
* Subjects who are breast-feeding.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects arriving for a mammography or breast ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05 (Estimated); Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel